CLINICAL TRIAL: NCT02874781
Title: Sublingual Microcirculation Data of Patients With Kidney Transplant
Brief Title: Microcirculation of Patients With Kidney Transplant
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201605035RINC
Record Dates: First submitted 2016-08-05; First posted 2016-08-22 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Microcirculation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study measures the sublingual microcirculation of patients with kidney transplant using MicroScan. The data will be compared with data of health volunteers and end stage renal disease patients on hemodialysis.

DETAILED DESCRIPTION:
This study measures the sublingual microcirculation of patients with kidney transplant using MicroScan. The data will be compared with data of health volunteers and end stage renal disease patients on hemodialysis. The microcirculation date includes total small vessel density, perfused small vessel density, proportion of perfused vessels, microvascular flow index, and heterogeneity index.

ELIGIBILITY:
Inclusion Criteria:

* patients with kidney transplant for more than one month

Exclusion Criteria:

* Body mass index (BMI) < 18.5 or > 30
* diagnosis of sepsis or trauma, or admitted to intensive care unit within one month before enrollment
* body temperature < 35.5 or > 37.5 Celsius
* patients with tongue resection
* non-native speaker

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with kidney transplant
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Total small vessel density | 6 hours
Perfused small vessel density | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No